CLINICAL TRIAL: NCT03009188
Title: Genetic Findings in a Chinese Family With Axenfeld-Rieger Syndrom
Status: Completed | Type: Observational
Sponsor: Aier Eye Hospital, Changsha (Other)
Responsible Party: Principal Investigator, Kuanshu Li, MD-candidate, Aier Eye Hospital, Changsha
Other Study IDs: AierEYC
Record Dates: First submitted 2016-12-31; First posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Genetic Findings in a Chinese Family With ARS
Keywords: Axenfeld-Rieger syndrom, genetic findings

STUDY DESIGN:
Observational Model: Family Based
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pedigree of the family with ARS: Nine members of the same family with ARS

SUMMARY:
Axenfeld-Rieger syndrome (ARS) is a rare autosomal dominant disorder, characterized by anterior segment abnormalities and systemic abnormalities. To date,two major genes, forkhead box C1 (FOXC1) on chromosome 6p25 and pituitary homeobox 2 (PITX2) on chromosome 4q25, have been demonstrated to cause ARS. In this study, we performed complete ophthalmologic examinations and analysis of FOXC1 and PITX2 of a Chinese family with ARS.

DETAILED DESCRIPTION:
Two genetions of a Chinese family with ARS were recruited to Aier Eye Hospital of Changsha.

Clinical evaluations: We performed full ophthalmologic examinations of all subjects, including: visual acuity, intraocular pressure measurements (Goldman), slit lamp, anterior segment photography, visual field test (Humphrey 750, Carl Zeiss, Germany), Anterior segment OCT (Carl Zeiss, Germany). If the refractive medium is clear, we also performed funduscopy, gonioscopic and retinal nerve fiber layer (RNFL) thickness measurements (Carl Zeiss, Germany).

Mutation analysis: About 2 ml of venous blood sampled from each subject and collected in Vacutainer tubes (Sanjiu Medical Technology Co., Ltd., Liuyang, China) containing EDTA. Genomic DNA was extracted from each blood using a genomic DNA mini kit for blood (Life Technologies), All coding exons, with flanking intronic regions, of FOXC1 and PITX2 were amplified using PCR with primers. The amplifed DNA was purifed by agarose gel electrophoresis and sequenced on a 3730/3700xl automated DNA sequencer (Applied Biosystems).

ELIGIBILITY:
Inclusion Criteria:

* a Chinese family with ARS

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Nine members of two genetions of a Chinese family with ARS
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2016-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Novel genetic findings in a Chinese family with Axenfeld-Rieger syndrom | Dec 1, 2016

IPD SHARING:
Plan to Share IPD: No